CLINICAL TRIAL: NCT06811519
Title: AI-based Prediction of Cardiac Function Using Echocardiography and Body Composition Data (ECHO-FIT Study)
Acronym: ECHO-FIT
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, In Hyun Jung, Professor, Yonsei University
Other Study IDs: ECHO-FIT
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Left Ventricular (LV) Systolic Dysfunction; Body Composition Measurement; Artificial Intelligence (AI)
Keywords: heart failure; left ventricular systolic dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic Test: Scanning body composition analyzer and performing AI algorithms: Diagnostic Test: Scanning body composition analyzer and performing AI algorithms
  Interventions: Diagnostic Test: Body Composition Analyzer (ACCUNIQ BC720)

INTERVENTIONS:
Diagnostic Test: Body Composition Analyzer (ACCUNIQ BC720) — Body Composition Analyzer (ACCUNIQ BC720)

SUMMARY:
This prospective observational study (ECHO-FIT Study) aims to develop and validate a predictive model for cardiac function, particularly left ventricular ejection fraction (LVEF), by integrating echocardiographic measurements with body composition data obtained from the QCCUNIQ BC 720 device.

The study plans to enroll 2,000 adult participants, comprising 1,000 individuals with normal LVEF (≥50%) and 1,000 with heart failure (LVEF <50%), all of whom will undergo standard-of-care echocardiography and body composition analysis.

By analyzing the relationships between key echocardiographic parameters (such as LVEF and diastolic function) and body composition measures (including fat mass, skeletal muscle mass, and total body water), we will develop a non-invasive prediction model capable of identifying individuals at higher risk of cardiac dysfunction.

This innovative approach has the potential to enhance early detection and personalized management of heart failure, reduce dependence on resource-intensive diagnostic procedures, and ultimately improve patient outcomes.

DETAILED DESCRIPTION:
Background and Rationale:

Heart failure represents a significant global health burden, characterized by high morbidity and mortality rates. While echocardiography remains the gold standard for heart failure diagnosis and monitoring, providing crucial measurements like left ventricular ejection fraction (LVEF) and diastolic function assessment, its widespread implementation is limited by resource constraints and operator dependency. Bioelectrical impedance analysis (BIA) offers a promising complementary approach, providing rapid and non-invasive assessment of body composition parameters that have shown correlations with cardiovascular outcomes. This study seeks to leverage the potential synergy between echocardiographic findings and body composition data to develop a more accessible screening tool for cardiac dysfunction.

Study Objectives:

* Primary: To develop and validate a predictive model for left ventricular function by integrating body composition data from the QCCUNIQ BC 720 device with standard echocardiographic parameters.
* Secondary:

  * To investigate correlations between body composition indices and echocardiographic measurements
  * To evaluate the utility of body composition analysis in identifying high-risk cardiovascular patients
  * To assess the model's potential as a screening tool in resource-limited settings

Methodology:

This single-center, prospective observational study will enroll 2,000 adults (≥20 years) undergoing routine echocardiography, equally divided between those with normal cardiac function (LVEF ≥50%) and heart failure (LVEF <50%). Participants will undergo body composition analysis using the QCCUNIQ BC 720 device within one week of their echocardiogram.

Data Collection and Analysis:

Comprehensive data collection will include standard echocardiographic parameters (LVEF, diastolic function, structural measurements) and detailed body composition analysis (fat mass, skeletal muscle mass, total body water). Statistical analysis will employ both traditional regression methods and advanced machine learning algorithms to develop the predictive model. Model validation will utilize k-fold cross-validation, with performance assessed through standard metrics including sensitivity, specificity, and area under the curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older.
* Undergoing a standard echocardiographic examination.
* Providing consent to undergo body composition analysis.
* Signing the informed consent form to voluntarily participate in the study.

Exclusion Criteria:

* Having a physical or mental condition that makes it impossible to conduct an echocardiogram or perform body composition analysis.
* Deemed inappropriate for study participation by the researcher (e.g., unable to cooperate).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is conducted in patients who have undergone transthoracic echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction < 50% | within 1 week
  Prediction of Left Ventricular Ejection Fraction < 50%

CONTACTS AND LOCATIONS:
Overall Officials: In Hyun Jung, MD., PhD., Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided